CLINICAL TRIAL: NCT03936582
Title: Promoting Small Business Support of Youth Physical Activity in Low-income, Minority Neighborhoods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Richard Suminski, Associate Professor, University of Delaware
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: BHAN32214719000
Record Dates: First submitted 2019-05-01; First posted 2019-05-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): All owners/managers of small businesses in 10 treatment neighborhoods will receive a request to support youth physical activity. The owners/managers will be able to direct support to specific programs, get recognized for their support, receive added information on the benefits of supporting such programs, have the oversight of an advisory board and interface with a local program representative
  Interventions: Behavioral: Treatment
- control (Active Comparator): All owners/managers of small businesses in 10 control neighborhoods will will receive a request to support youth physical activity. None of the other components of the treatment arm (e.g., direct support to specific programs, advisory board) will be provided.
  Interventions: Behavioral: Treatment

INTERVENTIONS:
Behavioral: Treatment — information already included in arm/group descriptions

SUMMARY:
An unacceptably high percentage of our nation's low-income, minority youth (< 18 years of age) are not regularly physically active. This contributes to extreme health disparities such as obesity rates nearly two-fold higher than those seen in white youth and greater risk for diabetes and related cardiometabolic disorders. The presence of quality youth physical activity opportunities (YPAO) enables and encourages physically active lifestyles. Unfortunately, quality YPAOs often are lacking in places where minority youth live, resulting in low activity levels and subsequent health issues that represent significant disparities in our society. The investigators' previous research found that small businesses (< 500 employees), which represent over 99% of all employers, are powerful resources for creating and improving YPAOs. In accordance with the Socioecological Model and established philanthropic principles, the investigators developed an alpha version of an intervention (alpha-i) for increasing small businesses' involvement with YPAOs. The investigators are now poised to create a beta version (beta-i) and conduct a pilot study of its impact on small business support for YPAOs and YPAO utilization by youth in low-income, minority neighborhoods. To meet this objective, the investigators will complete the following specific aims. Aim 1: Refine alpha-i components by completing focus groups with small business owners, YPAO providers, and parents/guardians of youth from low-income, predominantly minority neighborhoods. Results of the qualitative analysis will inform final tailoring of the intervention to create the beta-i which will be tested in Aim 2. Aim 2: Determine the effect of the beta-i on small business support for YPAOs in low-income, minority neighborhoods by conducting a plot cluster randomized-control trial with randomization at the neighborhood level. Intervention neighborhoods (n=10) will receive the beta-i while control neighborhoods (n=10) will be provided a standard practice intervention for a period of one year. The primary outcome for aim 2 will be the percentage of small businesses not supporting YPAOs at baseline that subsequently provide support for YPAOs at follow-up. The investigators also will consider the U.S. dollar equivalent of all types of support (monetary, goods/services and time) donated for YPAOs by small businesses. Aim 3: Examine the impact of the increased small business support for YPAOs on YPAO utilization by youth. The primary outcome will be the percent change in the number of youth participating in YPAOs from baseline and follow-up in the treatment and control neighborhoods. The proposed study is significant because it will provide evidence that an easily replicated approach can be used to increase small business support for YPAOs and that this support results in greater use of the YPAOs by youth. The investigators' next step will be to determine if YPAO changes resulting from increased small business support positively influence youth physical activity levels as measured by accelerometry. The investigators long-term goals are to create a nationally implementable practice for increasing support for YPAOs and strengthen the science of addressing health disparities in socially disadvantaged populations.

ELIGIBILITY:
Inclusion Criteria:

* small business (< 500 employees) in one of the 20 study areas with a physical, non-residential location.

Exclusion Criteria:

* large businesses (500 or more employees) not in one of the 20 study areas, does not have a physical location or the physical location is residential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
percentages of business supporting youth physical activity programs before and after intervention | one year
  Based on baseline and post-intervention survey data as well as information tracked on the project's websites.

SECONDARY OUTCOMES:
Youth physical activity utilization | one year
  Percent change in the number of youth participating in youth activity programs from baseline and follow-up in the treatment and control neighborhoods

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Yes
Project investigators will develop policies/procedures for sharing data with other interested parties not affiliated with the original project. These policies/procedures will be defined in a data-sharing agreement. The investigators will make the data and associated documentation available to users only under the data-sharing agreement that will provide for: a commitment to using the data only for research purposes and not to identify any individual participant/community by name, a commitment to securing the data using appropriate computer technology, determining the quality of the research proposal (significance, innovativeness, approach, and community benefit), a comprehensive dissemination plan (to community and scientific audiences), sharing of administrative costs to prepare data and related documentation, appropriate approvals of research protocols by the IRB and a commitment to destroying or returning the data after analyses are completed.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: after August 2020 for a period of 10 years
Access Criteria: see above

REFERENCES:
- [Derived] Suminski RR Jr, Robson S, Turner J, Plautz E. Promoting Small Business Support of Youth Physical Activity in Low-Income, Minority Neighborhoods: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Jul 30;8(7):e13141. doi: 10.2196/13141. PMID 31364602